CLINICAL TRIAL: NCT00549588
Title: The Efficacy of a Sunscreen With SPF30 and a After-sun-lotion in the Prevention of Polymorphic Light Eruption
Brief Title: Sunscreen and After-sun-lotion Protection in Polymorphic Light Eruption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Peter Wolf, MD, Principal Investigator, Medical University of Graz, Austria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 14-058 ex 03/04
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Polymorphic Light Eruption
Keywords: Polymorphic light eruption; UV radiation; photoprotection; sunscreen; DNA repair enzymes; after-sun-lotion
MeSH Terms: interventions — DNA Repair Enzymes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: After-sun-lotion with DNA repair enzymes — 2 mg/cm2 immediately after UV exposure
  Other Names: Proprietary after-sun lotion (Ateia Inc.)
Other: SPF30 sunscreen — 2 mg/cm2 2o min before UV exposure
  Other Names: SPF30 sunscreen (Ateia Inc.)
Other: Placebo after-sun-lotion — 2mg/cm2 immediately after UV exposure
  Other Names: Proprietary after sun lotion vehicle (Ateia Inc.)
Other: Intervention: none (only UV)

SUMMARY:
Polymorphic light eruption (PLE) is a common photodermatosis characterized by the appearance of itching, erythema, papules or vesicles on sun-exposed skin. Though etiology is unclear it is hypothesized that it is an abnormal immune response to autologous antigens generated by ultraviolet radiation (UVR). This randomized, double blinded left-right body side experimental comparison study was designed to assess the preventive effect of a sunscreen and topical DNA repair enzyme-containing after-sun lotion in PLE.

DETAILED DESCRIPTION:
A SPF 30 sunscreen (containing chemical and physical UV filters), an after-sun lotion containing liposomal encapsulated micrococcus luteus lysate with endonuclease activity and photolyase (active AS), and an after-sun placebo formulation (containing no DNA repair enzymes) (placebo AS) has been used in this study. Fourteen PLE patients were enrolled. On day 1, the individual minimal erythema dose (MED) was assessed on patients' buttock skin by exposure to a test ladder of solar-simulated UVR (xenon arc source, Oriel Corp. Darmstadt, Germany). From day 2 to 5, 0.75 individual MED exposures (increased by 0 to 25% per exposure, depending on the erythema response to a preceding dose) were given to a total of four 5-by-5 cm skin test fields on symmetrically located, individual PLE predilection sites on the trunk or extremities. The test fields were treated in randomized and double-blinded fashion either with SPF30 sunscreen 20 min before UVR exposure, active AS or placebo AS (all creams at a concentration of 2mg/cm2) immediately after UVR exposure, or left untreated. Sixty minutes after UVR exposure all test areas were treated with visible light (400 to 450nm, 5J/cm2) to activate the light dependent photolyase DNA repair mechanism. The photo test procedure led to the appearance of PLE symptoms in unprotected test fields of 12/14 (86%) patients, active AS-treated test fields of 6/14 (43%) patients (p<0.05), placebo AS-treated test fields of 10/14 (71%) patients (p, ns), and no (0%) sunscreen-protected test fields of any patient (p<0.0001 vs. unprotected test fields, Fisher exact test). These results provide evidence that i) DNA damage is a trigger of PLE, ii) increasing DNA repair can prevent induction of PLE symptoms, and iii) the use of sun care preparations containing DNA repair enzymes may be clinically useful for PLE patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PLE either by typical history and/or typical histology of lesions and/or positive phototesting results

Exclusion Criteria:

* Presence of or history of malignant skin tumors
* Dysplastic melanocytic nevus syndrome
* Photosensitive diseases such as porphyria, chronic actinic dermatitis, Xeroderma pigmentosum, basal cell nevus syndrome, and others
* Autoimmune disorders such as Lupus erythematosus or Dermatomyositis
* Psychiatric disorders
* Systemic treatment with steroids and/or other immunosuppressive drugs
* Pregnancy or lactation
* Antinuclear antibodies
* UV exposure in test fields within 8 weeks before study start
* General poor health status

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2004-02; Primary Completion 2004-06 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of symptoms of polymorphic light eruption | Prospective

SECONDARY OUTCOMES:
Pruritus | Prospective
Skin infiltration | prospective
Area affected | prospective
Erythema | prospective
Tanning | Prospective

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wolf, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Department of Dermatology, Graz, Austria